CLINICAL TRIAL: NCT06062589
Title: AK104 Combined With Iodine-125 Brachytherapy in the Treatment of Recurrent or Metastatic Cervical Cancer
Brief Title: AK104 Combined With I-125 Brachytherapy for Recurrent or Metastatic Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023109
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Iodine-125 particle brachytherapy — All enrolled patients' relapsed or metastatic lesions underwent image-guided radiation I-125 particle implantation brachytherapy (single implantation, half-life of 60 days, 99% of total dose given after 90 days). The prescribed dose is above 130Gy. Technical process: positioning and preoperative planning design; Template reset and particle implantation under the guidance of image system; Rapid and real-time intraoperative optimization; Postoperative dose validation.
Drug: AK104 — AK104 treatment (6mg/kg Q2W) starting within 1 week of particle implantation, for a total of 6 cycles or until disease progression, intolerable toxicity, investigator decision, withdrawal of informed consent, death, or other reasons as specified in the protocol.
  Other Names: Cadonilimab

SUMMARY:
The goal of this study is to determine efficacy and safety of AK104 combined with I-125 brachytherapy for recurrent or metastatic cervical cancer.

This is an open-label, single-center, observational study of AK104 with Iodine-125 brachytherapy in the treatment of recurrent or metastatic cervical cancer. 18 eligible patients will receive Iodine-125 brachytherapy (single implantation, half-life of 60 days, 99% of total dose given after 90 days), followed by AK104 treatment (6mg/kg Q2W) starting within 1 week of particle implantation, for a total of 6 cycles or until disease progression, intolerable toxicity, investigator decision, withdrawal of informed consent, death, or other reasons as specified in the protocol.

DETAILED DESCRIPTION:
Study Title AK104 combined with Iodine-125 brachytherapy in the Treatment of Recurrent or Metastatic Cervical Cancer

Study Objectives Primary Objective To explore the effectiveness of AK104 in combination with Iodine-125 brachytherapy in the treatment of recurrent or metastatic cervical cancer.

Secondary Objective To explore the safety of AK104 in combination with Iodine-125 brachytherapy in the treatment of recurrent or metastatic cervical cancer.

Study Endpoints Primary Endpoint Objective response rate (ORR) based on RECIST 1.1 evaluation.

Secondary Endpoints Disease control rate (DCR), progression-free survival (PFS), and 3-year overall survival rate (OS) based on RECIST 1.1 evaluation.

Safety assessment: Incidence and severity of adverse events (AE), clinically significant abnormal laboratory test results.

Target Population Patients with unresectable recurrent or metastatic cervical cancer who have undergone radical surgery and/or radical chemoradiotherapy and are suitable for local radiotherapy (non-central pelvic recurrence or oligometastasis in stage IVB).

Study Drug and Administration AK104, 6mg/kg Q2W, administered via intravenous infusion over 60 minutes (±10 minutes). For subjects unable to tolerate a 60-minute infusion, the infusion time may be extended up to 120 minutes. Dose adjustments are not allowed during treatment with AK104, but treatment may be delayed for a maximum of 12 weeks from the previous dose. Treatment will be discontinued if AK104 has been withheld for more than 12 weeks due to treatment-related immune-related adverse events (irAE) requiring corticosteroid therapy, or for reasons unrelated or potentially unrelated to AK104, but the investigator determines that the patient would benefit from continued treatment after discussion with the medical monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed cervical cancer, with recurrence or metastasis after previous systemic surgery, postoperative chemoradiotherapy, or radical chemoradiotherapy, and suitable for local radiotherapy (non-central pelvic recurrence or oligometastasis in stage IVB).
2. Pathologically and radiologically confirmed tumor with maximum diameter not exceeding the maximum diameter for particle treatment (5-7cm).
3. Age ≥18 years and ≤70 years, female at the time of signing the informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1, able to tolerate puncture.
5. Measurable lesions according to RECIST 1.1, with target lesions unsuitable for surgical treatment.
6. Expected survival time of more than 3 months.
7. Adequate organ function as per standard criteria for immunotherapy:

   * Absolute neutrophil count (ANC) ≥1.5×109/L
   * Platelets ≥75×109/L
   * Hemoglobin ≥90 g/L
   * Serum albumin ≥30 g/L
   * Total bilirubin (TBil) ≤1.5×ULN
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5×ULN; if there is liver metastasis, ALT and AST <5×ULN
   * Serum creatinine ≤1.5×ULN
   * Blood urea nitrogen (BUN) ≤2.5×ULN
   * Thyroid-stimulating hormone (TSH) ≤ upper limit of normal (ULN); if abnormal, investigate T3 and T4 levels, and if T3 and T4 levels are normal, the patient may be eligible.
8. Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days before starting study drug and agree to use a medically acceptable method of contraception during the study and for 3 months after the last dose of study drug.
9. Signed informed consent and the subject must understand the purpose of the study and the requirements for participation and voluntarily agree to participate.

Exclusion Criteria:

Potential subjects who meet any of the following criteria should be excluded from the study:

1. History of using anti-PD-1 antibodies, anti-CTLA-4 antibodies, TCR-T, CAR-T, or other immunotherapy within the past 4 weeks before the first dose, or participation in other anti-tumor drug clinical trials within the past 4 weeks before the first dose, or planned use of attenuated live vaccines during the study period.
2. Diagnosis of any other malignant tumor within the past 3 years.
3. Use the first dose, excluding intranasal and inhaled corticosteroids or physiologic doses of systemic corticosteroids (not exceeding 10 mg/day prednisolone or equivalent).
4. Patients with symptomatic, visceral metastasis, or short-term life-threatening complications risk, including uncontrollable large effusions (pleural, pericardial, or peritoneal), lymphangitis carcinomatosis, and 30% or more liver involvement.
5. Presence of any active autoimmune disease or history of autoimmune disease, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism. Patients with vitiligo or childhood asthma that has been completely resolved without any intervention during adulthood can be included. Patients with asthma requiring bronchodilators for medical intervention cannot be included.
6. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg despite optimal medical management).
7. Grade II or higher myocardial ischemia or myocardial infarction, uncontrolled arrhythmia (including QTc interval ≥450 ms for males or ≥470 ms for females), NYHA class III-IV heart failure, left ventricular ejection fraction (LVEF) <50% as determined by echocardiography. Patients who experienced myocardial infarction, New York Heart Association class II or higher heart failure, uncontrolled angina, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or acute ischemia or active conduction system abnormalities based on electrocardiogram within 6 months before enrollment.
8. Coagulation abnormalities (INR >1.5 or prothrombin time (PT) > upper limit of normal (ULN) + 4 seconds or APTT >1.5 ULN), bleeding tendency, or receiving thrombolysis or anticoagulation therapy.
9. Presence of obvious hemoptysis or expectoration of at least half a teaspoon (2.5 ml) of blood within 2 months before enrollment; or occurrence of significant clinically relevant bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, baseline occult blood++ in stool, or vasculitis within 3 months before enrollment; or occurrence of arterial/venous thromboembolic events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, or cerebral infarction), deep vein thrombosis, or pulmonary embolism within 6 months before enrollment.
10. Severe infection within 4 weeks before the first dose (e.g., requiring intravenous administration of antibiotics, antifungals, or antiviral agents), or unexplained fever >38.5°C during screening or within 4 weeks before the first dose.
11. History of substance abuse, inability to discontinue substance abuse or presence of psychiatric disorders.
12. Major surgery within 4 weeks before the first dose or presence of open wounds or fractures.
13. Factors significantly affecting oral drug absorption, such as inability to swallow, chronic diarrhea, or intestinal obstruction; or occurrence of fistula or perforation of hollow organs within 6 months.
14. Urinalysis showing urine protein ≥++, or confirmed 24-hour urine protein ≥1.0 g.
15. Human immunodeficiency virus (HIV) infection or known acquired immune deficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥500 IU/ml), hepatitis C (positive HCV antibodies and HCV-RNA above the detection limit of the assay), or concurrent infection with both hepatitis B and hepatitis C.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable recurrent or metastatic cervical cancer who have undergone radical surgery and/or radical chemoradiotherapy and are suitable for local radiotherapy (non-central pelvic recurrence or oligometastasis in stage IVB).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-10-11 (Estimated); Primary Completion 2025-01-11 (Estimated); Study Completion 2027-10-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From Baseline to 3 months
  ORR was assessed by the site Investigator using RECIST 1.1 and was defined as the percentage of patients with a confirmed overall response of CR or PR

SECONDARY OUTCOMES:
Disease control rate (DCR) | From Baseline to 2 years]
  DCR was assessed by the site Investigator using RECIST 1.1 and was defined as the percentage of patients with a confirmed overall response of CR or PR or SD.
Progression-free survival (PFS) | From Baseline to 2 years]
  the time of all participants from the start of the treatment to tumor progression
Overall survival rate (OS) | : From Baseline to 3 years]
  the time from the start of the treatment to the death of any cause.
The adverse events | From Baseline to 2 years
  The adverse events according to NCI-CTCAE v5.0